CLINICAL TRIAL: NCT02201381
Title: A Non Randomised, Non Blinded Real World Trial of the Safety, Tolerability and Effectiveness of Metabolic Medicines for the Treatment of Cancer Compared Against Matched Controls
Brief Title: Study of the Safety, Tolerability and Efficacy of Metabolic Combination Treatments on Cancer
Acronym: METRICS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Prospective recruitment not possible
Sponsor: Health Clinics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Metabolic Cancer 001
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cancer; Overall Survival
Keywords: Cancer; Cancer Treatments; Cancer Palliative Care; Metabolic; Metabolism; Existing Medicines; Licensed Medicines; Real World; Breast Cancer; Triple Negative Breast Cancer; Colon Cancer; Prostrate Cancer; Brain Cancer; Ovarian Cancer; Pancreatic Cancer; AML; CML; Leukemea; Metformin; Statins; Mebendazole; Doxycycline; Ibuprofen; Metastatic
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms; Colonic Neoplasms; Brain Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Metformin; Atorvastatin; Doxycycline; Mebendazole

STUDY DESIGN:
Intervention Model Description: Matched historical control comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metabolic Treatment (Experimental): Subjects will take the following treatments and have their data collected from their medical records every 3 months.
  * Oral atorvastatin up to 80mg uid, for study duration.
  * Oral metformin up to 1000mg uid, increased to bid if tolerated after 2 weeks, for study duration.
  * Oral doxycycline 100mg uid, for study duration.
  * Oral Mebendazole 100mg uid, for study duration.
  Interventions: Drug: Metabolic treatment

INTERVENTIONS:
Drug: Metabolic treatment — While subjects are being treated with the four metabolic drugs, every 3 months they will bring in their medical records and data will be collected to determine the effect of the intervention
  Other Names: Metformin; Atorvastatin; Doxycycline; Mebendazole

SUMMARY:
The purpose of this study is to determine the effectiveness of a regimen of selected metabolic treatments for patients with cancer in a real world setting and to conduct exploratory analysis on the relationship between the degree of response and changes in biochemical markers (such as glucose and lipid levels).

DETAILED DESCRIPTION:
*This study has been designed to collect data prospectively and to retrospectively analyse data on the metabolic treatments within the cancer clinic. The retrospective study is ongoing, while the prospective study has not yet started.*

This is a real world study since this gives the best opportunity to properly examine the effect of multi-drug regimens in representative populations. Including a standard of care arm is inappropriate, in a population in which that standard of care has already been shown to be ineffective or intolerable.

Patients will be sent to the study clinic directly by their Health Care Professionals ("HCP's") .

The study will consist of a pre-screening visit to determine eligibility for inclusion into the study, an initiation visit and then a follow up visit every three months thereafter. If required, unscheduled visits may take place. Day 0 (baseline) for each patient will be the initiation visit when study treatment is started.

Prior to conducting any study-related procedures, subjects will provide written informed consent, eligibility will be assessed, a medical history and past medical records will be taken and vital signs will be measured. These records will include the stage of their disease, response to previous cancer therapy, their prior and current medications and any specific regimen they are currently on for their cancer. If prior medical records do not contain sufficient information to determine a baseline for the patient, additional blood tests and scans will be undertaken as appropriate.

Patients will be monitored quarterly thereafter when blood tests (e.g. safety parameters, glucose, cholesterol, immune response and cancer markers where applicable) and scans (where applicable) will be taken.

All patients will be on the same drug regimen (see below) at the same doses throughout the study. All patients will be followed up until they choose to leave the study, or death.

Data from all patients recruited to the study will be analysed using an Intention-to-treat (ITT) philosophy, so data will be included in the primary analysis irrespective of whether the dose regimen was followed throughout the study. If appropriate, and numbers allow, analysis will also be conducted on the Per Protocol population, comprising those patients who adhere to the regimen as prescribed.

Survival analysis methods will be used to estimate the Overall survival associated with the study regimen for each type of cancer. These estimates will be interpreted in the light of data obtained from the literature, and from eliciting expert opinion. Bayesian methods may be used where appropriate.

Tumour response, where applicable, will be summarised in tables and graphs. Estimates of response rates will be presented for each cancer type with confidence intervals.

The relationship between changes in biochemistry values (glucose, lipids) and efficacy outcomes (Progression Free Survival (PFS), Overall Survival (OS) and HRQoL) will be investigated graphically, or using other methods as appropriate.

Further exploratory analysis to investigate the effects of other factors such as age , ethnic backgrounds , cancer stage, and response to prior therapy, will also be conducted in order to try and characterise the profile of patients most likely to benefit from the study regimen.

The characteristics of patients on the regimen and those who do not stay on the regimen, for whatever reason, will be summarised to see whether there is any observed bias. If appropriate, methods will be used to adjust for any observed bias, for example using propensity scores. OS can then be assessed adjusted for this to try and mitigate for any possible risk of bias which can occur in uncontrolled studies. Furthermore, by enrolling all eligible patients over a specified time frame, it is hoped that the risk of bias should be further reduced. In addition, a large number of patients are expected to participate in the study.

ELIGIBILITY:
Inclusion criteria

1. Male or female 18-85 years old;
2. Diagnosed with cancer and have had such diagnosis confirmed by scan, blood markers and/or biopsy;
3. Is receiving or will shortly receive standard of care therapy or has completed standard of care treatment; and
4. Signed and dated written informed consent from the participant or LAR.

Exclusion Criteria:

1. Pregnant or lactating females or females who are planning a pregnancy during the course of the study;
2. Major organ failure, renal, lung and liver failure;
3. Participants having active liver disease or unexplained persistent elevation of serum transaminases > 3 times the upper limit of normal;
4. Participants with diabetic ketoacidosis or diabetic pre-coma;
5. Participants with a creatinine clearance < 60mL/min;
6. History of cardiac or respiratory failure;
7. History of recent myocardial infarction;
8. Ileum, colon or stomach part or full removal rendering them unable to take the study medicines;
9. Unable to eat or keep food or medicines down or is being fed intravenously;
10. Is too frail and weak to withstand the study medicines in the opinion of the study doctor;
11. Is Unlikely to survive more than 1 month under standard of care, in the opinion of the study doctor
12. Hypersensitivity to any of the treatment drugs or excipients;
13. If the patient is on any medicines contraindicated with the study medicines (see Appendix 3);
14. Mentally incapacitated and no guardian able to sign on patients Clinical study protocol, version 5.0 METRICS TRIAL, Metabolic Cancer 001 5th Apr 2016 Confidential Page 5 of 65 behalf;
15. History or presence of alcohol or substance abuse;
16. Participation in a clinical trial of an investigational medicinal product that is viewed by the Study Physician to be a significant risk to the participant's safety;
17. Direct employee of the study site.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 5 years
  Overall survival for all cancer types and for each cancer type (years and months)

SECONDARY OUTCOMES:
Change in primary tumour size cancer types and by cancer type. | up to 5 years
  Tumour size for all cancer types and for each cancer type. Units of size vary depending on cancer type.
Change in tumour spread (metastasis) | up to 5 years
  Tumour spread (metastasized) to other tissues/organs, for all cancer types and for each cancer type. This is measured as either 0 for no spread or 1 for confirmed spread.
Change in tumour number | up to 5 years
  Tumour number for all cancer types and for each cancer type
Change in cancer biomarkers (blood, urine or biopsy) | up to 5 years
  Cancer biomarkers for all cancer types and for each cancer type. Units of measurement vary depending on the cancer type. When biomarkers, either alone or in combination with other biomarkers, are raised above normal they are seen as predictive of cancer of progression. If returned to normal are indicative of treatment response.

OTHER OUTCOMES:
Incidence of treatment related adverse events | 5 years
  Adverse events reported by the subject or their HCP.
  • Quarterly assessment of routine laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Samir Agrawal, MRCP FRCPath, Principal Investigator — Care Oncology Clinic
Locations (1):
- Care Oncology Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No